CLINICAL TRIAL: NCT02833181
Title: Evaluation of Circadian Variation of EEG Using BIS Monitor in ICU Patients
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar do Tâmega e Sousa (Other)
Responsible Party: Principal Investigator, Mariana Marques da Cunha, MD, Centro Hospitalar do Tâmega e Sousa
Other Study IDs: BISEECS
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: EEG Circadian Variation of ICU Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Awake patients: Awake patients
  Interventions: Device: BIS monitor
- Sedated patients
  Interventions: Device: BIS monitor
- Sedated and curarized patients
  Interventions: Device: BIS monitor

INTERVENTIONS:
Device: BIS monitor — Monitoring circadian variation of EEG

SUMMARY:
The investigators propose to evaluate circadian variation of EEG using BIS (bispectral index) monitor in ICU patients in three different groups: non-sedated, only sedated and sedated and curarized. BIS monitor values as SR (suppression rate), SEF (Spectral edge frequency), bispectral index and EMG (electromyography) during 24 hours in admitted patients except acute neurological disease.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in the ICU
* Over 18 years old

Exclusion Criteria:

* Acute neurological disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Circadian EEG variation | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Tâmega e Sousa, Penafiel, Portugal